CLINICAL TRIAL: NCT00754598
Title: A Multicenter, Controlled Clinical Trial to Evaluate the Hologic 3-D Tomosynthesis Mammography System Used in Conjunction With Conventional 2-D Digital Mammography
Brief Title: Evaluation of a 3-D Tomosynthesis Mammography System Used in Conjunction With Conventional 2-D Digital Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Diagnostic
Other Study IDs: 05-01
Record Dates: First submitted 2008-09-10; First posted 2008-09-18 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; digital mammography; tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Tomosynthesis digital mammography imaging system — a full-field digital mammography system where multiple images are acquired at various angles near the normal to the detector. Breast compression is performed in a standard geometry. The acquired images are reconstructed using mathematical algorithms, not unlike CT reconstructions, to generate a set of thin slices parallel to the breast platform. The reconstructed slices can be viewed individually or in a movie format.
  Other Names: Genesis; Hologic Tomosynthesis; Tomo

SUMMARY:
This was a multi-center, prospective clinical trial in which the subject was her own control. Approximately 950-1400 female subjects were enrolled at five (5) sites in the United States. Subjects were from either a Screening population or a biopsy population and were imaged first on a conventional 2D full filed digital mammography system then on a 3D tomosynthesis system.

The resulting images from the this portion of the study were then randomized into a reader study.

The purpose of this clinical study was to compare the 3-D tomosynthesis system used in conjunction with a conventional 2-D digital imaging system (2-D plus 3-D images) to the conventional 2-D digital imaging system (2-D images), and to determine whether the 2-D plus 3-D images compared to the 2-D images alone would:

1. Reduce the recall rate And/or
2. Improve ROC area due to improved breast cancer detection and/or improved lesion classification.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Any ethnic origin
* No contraindication for screening mammography

Exclusion Criteria:

* Significant breast trauma
* Pregnancy
* Lactating
* Breast implants
* Previous breast cancer
* Previous surgical biopsy
* Placement of an internal breast marker
* Unable to understand and or execute written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1183 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To detect a 20% reduction in the recall rate when comparing the recall rate using the BIRADS 0 scores of the 2-D plus 3-D images to the 2-D images. | 10-12 months

SECONDARY OUTCOMES:
To detect a 0.05 increase in the area under the ROC curve when comparing 2-D plus 3-D images to the 2-D images. | 10-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rafferty, M.D, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Iowa Medical Center, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Magee Women's Hospital, Pittsburgh, Pennsylvania